CLINICAL TRIAL: NCT05987163
Title: A Randomized, Evaluator-blinded, Parallel Group, Comparator-controlled, Multicenter Study to Evaluate the Safety and Effectiveness of GP0116 for Correction of Moderate to Severe Dynamic Facial Wrinkles and Folds, Such as Nasolabial Folds.
Brief Title: Study to Evaluate the Safety and Effectiveness of GP0116
Acronym: NLF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 43N3US2204
Record Dates: First submitted 2023-04-04; First posted 2023-08-14 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Skin Manifestations
MeSH Terms: conditions — Skin Manifestations

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (2):
- GP0116 (Experimental)
  Interventions: Device: GP0116
- FDA Approved Device (Active Comparator)
  Interventions: Device: Active Comparator: FDA approved dermal filler device (RHA 3)

INTERVENTIONS:
Device: GP0116 — GP0116 is an injectable, sterile, transparent product.
  Arms: GP0116
Device: Active Comparator: FDA approved dermal filler device (RHA 3) — FDA approved dermal filler device (RHA 3)
  Arms: FDA Approved Device

SUMMARY:
This is a prospective, randomized, evaluator-blinded, comparator-controlled, parallel group, multicenter study in the U.S. for correction of moderate to severe dynamic facial wrinkles and folds, such as nasolabial folds (NLFs).

ELIGIBILITY:
Inclusion Criteria:

* Men and non-pregnant, non-breastfeeding women aged 22 years or older.
* WSRS grade of 3 or 4 (moderate to severe folds) on each NLF as assessed by the Blinded Evaluator. The WSRS for each NLF does not need to be equal.
* Intent to undergo treatment for correction of both left and right NLF.

Exclusion Criteria:

* Known/previous allergy or hypersensitivity to any injectable hyaluronic acid (HA) gel
* Known/previous allergy or hypersensitivity to local anesthetics
* Previous or present severe or multiple allergies manifested by severe reactions
* Previous facial surgery near the treatment area

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 186 (Estimated)
Dates: Start 2023-04-12 (Actual); Primary Completion 2024-10-29 (Actual); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
To demonstrate non-inferiority of GP0116 versus a comparator control | At 3 months after Baseline
  To demonstrate non-inferiority of GP0116 versus a comparator control in correction of NLFs by comparing change from baseline based on the Blinded Evaluator's live assessment of NLF correction at Month 3 using the Wrinkle Severity Rating Scale (WSRS).

CONTACTS AND LOCATIONS:
Locations (19):
- United States (18):
  - Galderma Investigational Site (Site#8074), Santa Monica, California
  - Galderma Investigational Site (Site#8478), Vista, California
  - Galderma Investigational Site (Site#8680), Westport, Connecticut
  - Galderma Investigational Site (Site#8479), Bradenton, Florida
  - Galderma Investigational Site (Site#7030), Coral Gables, Florida
  - Galderma Investigational Site (Site#8284), Coral Gables, Florida
  - Galderma Investigational Site (Site#8126), West Palm Beach, Florida
  - Galderma Investigational Site (Site#7042), Atlanta, Georgia
  - Galderma Investigational Site (Site#8580), New Orleans, Louisiana
  - Galderma Investigational Site (Site#8481), Chestnut Hill, Massachusetts
  - Galderma Investigational Site (Site#8631), Birmingham, Michigan
  - Galderma Investigational Site (Site#8658), New York, New York
  - Galderma Investigational Site (Site#8482), Chapel Hill, North Carolina
  - Galderma Investigational Site (Site#8648), Wilmington, North Carolina
  - Galderma Investigational Site (Site#8783), Cincinnati, Ohio
  - Galderma Investigational Site (Site#8496), Nashville, Tennessee
  - Galderma Investigational Site (Site#8662), Spring, Texas
  - Galderma Investigational Site (Site#7047), Arlington, Virginia
- Galderma Investigational Site (Site#8784), San Juan, Puerto Rico